CLINICAL TRIAL: NCT04847544
Title: A Randomized, Double-Blind, Placebo-Controlled, Clinical Trial to Evaluate the Safety, Tolerability, Efficacy, and Pharmacodynamics of ADX-629 Administered Orally for the Treatment of COVID-19
Brief Title: A Randomized, Double-Blind, Placebo-Controlled, Clinical Trial to Evaluate the Safety, Tolerability, Efficacy, and Pharmacodynamics for the Treatment of COVID-19.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aldeyra Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ADX-629-COVID-19-001
Record Dates: First submitted 2021-04-13; First posted 2021-04-19 (Actual); Results first posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2022-05

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — ADX-629

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ADX-629 300 mg administered orally twice daily (BID) for up to 28 days. (Experimental)
  Interventions: Drug: ADX-629
- Placebo administered orally BID for up to 28 days. (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ADX-629 — ADX-629 administered orally twice daily (BID) for up to 28 days.
  Arms: ADX-629 300 mg administered orally twice daily (BID) for up to 28 days.
Drug: Placebo — Placebo administered orally BID for up to 28 days.
  Arms: Placebo administered orally BID for up to 28 days.

SUMMARY:
A Randomized, Double-Blind, Placebo-Controlled, Clinical Trial to Evaluate the Safety, Tolerability, Efficacy, and Pharmacodynamics of ADX-629 Administered Orally for the Treatment of COVID-19

ELIGIBILITY:
Inclusion Criteria:

* Is a male or female greater than or equal to18 years of age at Screening;
* Is willing and able to sign and date (or has a legally authorized representative willing to sign and date) a written (or electronic) informed consent form or provide equivalent consent per Food and Drug Administration guidelines on COVID-19 clinical trials;
* Has a documented, laboratory-confirmed severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2) infection as determined by polymerase chain reaction, a SARS-CoV-2 antigen test, or another commercial or public health assay, within 3 days (72 hours) of randomization;
* Has COVID-19 of moderate severity, as defined by the following: Positive testing by standard reverse transcription polymerase chain reaction assay or equivalent testing; Symptoms of illness with COVID-19, which could include any of the following: cough, fever, shortness of breath, chest pain, abdominal pain, nausea/vomiting, diarrhea, body aches, weakness/fatigue, or new loss of taste or smell; Clinical signs suggestive of illness with COVID-19, such as respiratory rate greater than or equal to 20 breaths per minute, saturation of oxygen greater than 93% on room air at sea level, or heart rate greater than or equal to 90 beats per minute; and No clinical signs indicative of severe or critical severity.

Exclusion Criteria:

* Has an NIAID ordinal scale score <5;
* Is on high-flow oxygen or any form of noninvasive ventilation, excluding continuous positive airway pressure (CPAP) alone for sleep disorders (e.g., obstructive sleep apnea);
* Has significant cardiovascular disease, defined by myocardial infarction, arterial thromboembolism, or cerebrovascular thromboembolism within 3 months prior to randomization; symptomatic dysrhythmias or unstable dysrhythmias requiring medical therapy; angina requiring therapy; symptomatic peripheral vascular disease; New York Heart Association Class 3 or 4 congestive heart failure; Grade 3 hypertension (diastolic blood pressure greater than or equal to 100 mmHg or systolic blood pressure greater than or equal to 160 mmHg); history of congenital prolonged QT syndrome, or known dyslipidemia;
* Is currently taking any investigational products, other than the study drug;
* Has any other condition that, in the opinion of the Investigator, could interfere with (or for which the treatment might interfere with) the conduct of the clinical trial or interpretation of the clinical trial results or that would place the subject at undue risk by participating in the clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-03-31 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2021-10-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Research Center of Miami II, Inc., Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- ADX-629: ADX-629 300 mg administered orally twice daily (BID) for 28 days
- Placebo: Placebo administered orally BID for 28 days
Period: Overall Study
Arm/Group | ADX-629 | Placebo
Started | 7 | 4
Completed | 7 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- ADX-629: ADX-629 300 mg administered orally BID for 28 days
- Total: Total of all reporting groups
Arm/Group | ADX-629 | Placebo | Total
Number analyzed (Participants) | 7 | 4 | 11
Age, Continuous [Mean (Full Range); unit: years] | 49.0 [30 to 67] | 55.3 [50 to 61] | 51.3 [30 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 4 | 2 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 7
  Not Hispanic or Latino | 3 | 1 | 4
SARS-CoV-2 Test Severity [Count of Participants; unit: Participants]
  SARS-CoV-2 Infection without Symptoms | 0 | 0 | 0
  Mild COVID-19 | 2 | 1 | 3
  Moderate COVID-19 | 5 | 3 | 8
  Severe COVID-19 | 0 | 0 | 0
  Critical COVID-19 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Serious Adverse Events
Description: Safety was assessed through serious adverse event reporting.
Time Frame: The safety assessment period was Days 1 - 28.
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | ADX-629 | Placebo
Number analyzed (Participants) | 7 | 4
Participants | 0 | 1

2. Secondary Outcome: Change From Baseline in the National Institute of Allergy and Infectious Diseases (NIAID) Scale
Description: Change from baseline in the National Institute of Allergy and Infectious Diseases (NIAID) scale, which is an eight-point ordinal scale (1 = death, 8 = not hospitalized with no limitation of activities) where a lower score indicates more severity. The least squares mean (standard error) was derived from mixed model repeated measures which included change from baseline as the response variable, treatment, day of visit, treatment-by-visit interaction as fixed effects, and baseline as a covariate.
Time Frame: The efficacy assessment period was 4 weeks; baseline was defined as Day 1 prior to first dose.
Population: Intent-to-treat population with last observation carried forward (LOCF)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | ADX-629 | Placebo
Number analyzed (Participants) | 7 | 4
score on a scale | 0.86 (0.366) | 0 (0.484)

ADVERSE EVENTS:
Time Frame: The period of time over which adverse events were collected was approximately 28 days.
Arm/Group | ADX-629 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/7 | 1/4
Other Adverse Events (participants affected / at risk) | 2/7 | 1/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ADX-629 (N=7) | Placebo (N=4)
COVID-19 with hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ADX-629 (N=7) | Placebo (N=4)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Elevated Alanine Aminotransferase (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-12-11): https://cdn.clinicaltrials.gov/large-docs/44/NCT04847544/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-18): https://cdn.clinicaltrials.gov/large-docs/44/NCT04847544/SAP_001.pdf